CLINICAL TRIAL: NCT00536042
Title: Open-Label Trial of the Use of Minocycline as an Anti-Inflammatory Agent in the Treatment of Asthma
Brief Title: Open-Label Trial of the Use of Minocycline in the Treatment of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Rauno Joks, MD, Associate Professor of Clinical Medicine, State University of New York - Downstate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: open mino
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: minocycline; asthma; oral steroids; IgE
MeSH Terms: conditions — Asthma; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- minocycline (Experimental): addition of minocycline to standard asthma care as add-on therapy: 150 mg bid to 250 mg bid for up to one year
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — addition of 150 mg to 250 mg po bid to standard asthma care regiment
  Other Names: Minocin

SUMMARY:
The tetracycline minocycline has, in addition to its anti-infective properties, anti-inflammatory properties which may be of use in the treatment of asthma. This study evaluates the benefit of minocycline as add-on therapy for adults with asthma.

DETAILED DESCRIPTION:
Adult asthmatic (ages 18 to 75 years) with a history of moderate to severe persistent asthma are given minocycline capsules as add-on therapy for treatment of asthma. Treatment is for one year. Dosing begins at 150 mg twice daily and can increase every eight weeks by 50mg BID to a maximum of 250 mg twice daily. This is as per patient tolerance as minocycline can cause dizziness and stomach upset, as well as effects of liver enzymes.Patients undergo routine blood toxicity screens every two months, at which time spirometry is performed Exclusion criteria: pregnant women (adequate contraception in mandated) previous history of hypersensitivity to tetracyclines, chronic liver disease Outcome measures: improvement in FEV1 and other spirometric parameters, decrease in oral steroid requirements, change in total serum IgE, improvement in quality of life

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 to 75 yrs)
* Mild to severe asthma
* History of or current oral steroid use to control asthma atopy

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1997-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Improvement in FEV1 on spirometry | one year

SECONDARY OUTCOMES:
decrease in total serum IgE | one year
decrease in oral steroid requirements | one year
improvement in quality of life scores | one year

CONTACTS AND LOCATIONS:
Overall Officials: Rauno Joks, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided